CLINICAL TRIAL: NCT00721344
Title: A Phase 1, Randomized, Double-Blind, Cross-Over, Placebo- and Active-Controlled Cardiac Safety Study of Therapeutic and Supratherapeutic Doses of Fumaryl Diketopiperazine Administered as Technosphere® Inhalation Powder in Healthy Subjects
Brief Title: A Study to Determine if Technosphere® Inhalation Powder (FDKP) Causes ECG Changes (QTc) Following the Medication's Inhaled Administration.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MKC-T-131
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Subjects
Keywords: Healthy males and females
MeSH Terms: interventions — 3,6-bis(N-fumaryl-N(n-butyl)amino)-2,5-diketopiperazine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Technosphere Inhalation Powder (FDKP); Drug: Moxifloxacin; Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Technosphere Inhalation Powder (FDKP); Drug: Moxifloxacin; Drug: Placebo
- 3 (Experimental)
  Interventions: Drug: Technosphere Inhalation Powder (FDKP); Drug: Moxifloxacin; Drug: Placebo
- 4 (Experimental)
  Interventions: Drug: Technosphere Inhalation Powder (FDKP); Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: Technosphere Inhalation Powder (FDKP) — Technosphere® Inhalation Powder 20mg
Drug: Moxifloxacin — Tablets 400mg
Drug: Technosphere Inhalation Powder (FDKP) — Technosphere® Inhalation Powder 40mg
Drug: Placebo — Placebo cartridges

SUMMARY:
48 healthy adult male & female subjects will be enrolled in this study to determine the effect of Technosphere® Inhalation Powder (FDKP) on the QT interval of the EKG. Eligible subjects will be randomized into a dosing regimen after admission.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, cross-over, placebo- and active-controlled cardiac safety study in 48 healthy subjects (both male and female subjects) designed to assess the effect of FDKP on cardiac repolarization, if any, following introduction of Technosphere® Inhalation Powder via inhalation. Each trial subject will be administered 20 mg of FDKP, 40 mg of FDKP, 400 mg oral dose of moxifloxacin (active), and placebo in a crossover design during an 11 day in-patient stay.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary Function Tests (PFTs) results within study specified limits.
* Female subjects of childbearing potential must be non-pregnant and non-lactating and have a negative serum pregnancy test prior to enrollment into the trial.
* Body Mass Index = 19 and = 30 kg/m2
* Absence of recent drug or alcohol abuse
* Able to provide written informed consent, follow study procedures and remain in-patient for the entire treatment period
* Non-smoking (> 6 months)

Exclusion Criteria:

* History of significant renal, pulmonary, rheumatological, hematological, neurological or psychiatrics disorder
* Clinically significant major organ disease
* Evidence or history of clinically significant allergies (except for untreated, asymptomatic, seasonal allergies at time of dosing);
* Current or previous chemotherapy or radiation therapy that could cause lung toxicity
* History of diabetes or taking any medications to treat diabetes
* Clinically significant abnormal findings on physical exam, ECG, vital signs, clinical laboratory testing and medical history
* Hypokalemia (calcium below lower limit of normal).
* Previous exposure to Technosphere® Inhalation Powder
* Participation in another clinical trial of an investigational drug or device within 30 days prior to Visit 3
* Significantly excessive consumption of food or beverages with xanthine or caffeine
* Unwilling to avoid alcohol 48 hours prior to study enrollment and during study
* Unwilling to avoid strenuous activity for 48 hours prior to study enrollment and during study
* Positive HIV or Hepatitis test
* Any acute illness or fever within 72 hours of study dosing
* Medication use (with exception of acetaminophen and hormonal birth control) or herbal use within 7 days of Visit 2
* Unwillingness to remain in a quiet, controlled environment (i.e., no TV, music, games, etc during specific timepoints) or unwilling to remain supine during specific timepoints
* Unwillingness to consume a study-specific diet
* Blood donation within 8 weeks prior to Visit 2
* History of chronic obstructive pulmonary disease (COPD), clinically proven asthma and/or any other clinically important pulmonary disease confirmed by pulmonary function testing and/or radiological finding
* Active respiratory infection or persistent symptoms of such infection
* History of risk factors for Torsades de pointes (TdP) [e.g., heart failure, hypokalemia, family history (parents or siblings) of Long QT Syndrome], history of fainting, unexplained loss of consciousness or convulsions
* History of cardiac arrhythmia, of taking anti-arrhythmia drugs, significant cardiovascular dysfunction, myocardial dysfunction, cardiac surgery, transient attacks of ischemia or cerebrovascular accidents
* An abnormal screening ECG which is interpreted by the Clinical Site Investigator to be clinically significant
* Sustained supine resting systolic blood pressure > 140 mm Hg or < 100 mm Hg and /or diastolic blood pressure >95 mm Hg at study entry Baseline pulse rate of < 45 beats per minute or > 100 beats per minute

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the time-matched, placebo-subtracted change from baseline in QTc after a supratherapeutic dose of Technosphere Inhalation Powder | 11 days

SECONDARY OUTCOMES:
The time-matched change from baseline in QTc after therapeutic dose Technosphere® Inhalation Powder based on an individual correction (QTcI) method. | 11 days
The maximum change in time-matched, placebo-subtracted QT interval corrected by Fridericia formula (QTcF) and Bazett formula (QTcB), respectively, for supratherapeutic dose of Technosphere® Inhalation Powder. | 11 Days
The maximum change in time-matched, placebo-subtracted QT/QTc intervals by Fridericia formula (QTcF), and by Bazett formula (QTcB), respectively, for therapeutic dose of Technosphere® Inhalation Powder. | 11 Days
Change in ECG morphological patterns | 11 Days
Heart rate and RR interval. | 11 Days
PR interval. | 11 Days
QRS interval. | 11 Days
Correlation between the QTcI change from baseline and plasma concentrations of FDKP. | 11 Days
Plasma concentrations of FDKP. | 11 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Charles River Clinical Services Northwest, Tacoma, Washington, United States